CLINICAL TRIAL: NCT01896505
Title: An Open-Label Phase IB Trial To Evaluate the Effects of Food and Formulation on Pharmacokinetics of the Oral Selective Inhibitor of Nuclear Export/SINE Compound KPT-330 in Patients With Soft-Tissue or Bone Sarcoma
Brief Title: A Phase I Trial to Assess the Effects of Food and Formulation on PK of KPT-330 in Patients With Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-003
Record Dates: First submitted 2013-06-11; First posted 2013-07-11 (Estimated); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Sarcoma
Keywords: Bone sarcoma; Soft-tissue sarcoma; Sarcoma; KPT-330; Food; Effects; Selinexor
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 30 milligrams per meter square (mg/m^2) orally twice weekly in treatment sequence ABCD (Treatment A: fasted, tablet formulation on Day 1 of Week 1; Treatment B: high-fat meal, tablet formulation on Day 1 of Week 2; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 3; Treatment D: low-fat meal, capsule formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
  Interventions: Drug: KCP-330
- Arm 2 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence BADC (Treatment B: high-fat meal, tablet formulation on Day 1 of Week 1; Treatment A: fasted, tablet formulation on Day 1 of Week 2; Treatment D: low fat meal, capsule formulation on Day 1 of Week 3; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
  Interventions: Drug: KCP-330
- Arm 3 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 50 mg/m^2 first generation tablets twice weekly on Days 1 and 3 of each week within 30 minutes of solid food consumption.
  Interventions: Drug: KCP-330
- Arm 4 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 60 mg/m^2 orally in treatment sequence ABC (Treatment A: current [1st generation] tablets on Day 1 of Week 1; Treatment B: new [2nd generation] tablets on Day 1 of Week 2; Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
  Interventions: Drug: KCP-330
- Arm 5 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 60 mg/m^2 orally in treatment sequence CAB (Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 1; Treatment A: current [1st generation] tablets on Day 1 of Week 2; Treatment B: new [2nd generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
  Interventions: Drug: KCP-330
- Arm 6 (Experimental): Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 60 mg/m^2 orally in treatment sequence BCA (Treatment B: new [2nd generation] tablets on Day 1 of Week 1; Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 2; Treatment A: current [1st generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
  Interventions: Drug: KCP-330

INTERVENTIONS:
Drug: KCP-330
  Other Names: Selinexor

SUMMARY:
The purpose of this research study is to find out more information such as: to determine the effects of high and low fat foods on the pharmacokinetics (PK) of oral KPT-330 tablets and to compare PK of capsules and tablets in Arms 1 and 2; to evaluate tumor response in sarcoma participants in Arm 3; to compare the PK of 60 milligrams (mg) of the new, 2nd generation tablet formulation and 60 mg of the selinexor suspension formula to the current, 1st generation tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed soft tissue or bone/cartilage sarcoma. Patients with sarcoma of small round blue cell tumor types are allowed. Gastrointestinal stromal tumors (GIST) are excluded.
2. Patients must have received at least one prior anticancer regimen for metastatic disease unless there is no other therapy available and evidence of progressive disease on study entry. Patients with stable disease will be included if there has been failure to respond to another drug(s) within the previous 3 months

Exclusion Criteria:

1. Patients with known liver metastases
2. Radiation, chemotherapy, immunotherapy, any other systemic anticancer therapy or participation in an investigational anti-cancer study ≤ 3 weeks prior to initiation of therapy
3. Patients with known brain metastasis
4. Patients with any gastrointestinal dysfunctions that could interfere with the interpretation of the food effect data
5. Patients with known intolerance to low or high fat meals
6. In the opinion of the investigator, patients who are significantly below their ideal body weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kauffman, MD, Ph.D, Study Director — Karyopharm Therapeutics Inc
Locations (2):
- Memorial Sloan Kettering Cancer Centre, New York, New York, United States
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gounder MM, Zer A, Tap WD, Salah S, Dickson MA, Gupta AA, Keohan ML, Loong HH, D'Angelo SP, Baker S, Condy M, Nyquist-Schultz K, Tanner L, Erinjeri JP, Jasmine FH, Friedlander S, Carlson R, Unger TJ, Saint-Martin JR, Rashal T, Ellis J, Kauffman M, Shacham S, Schwartz GK, Abdul Razak AR. Phase IB Study of Selinexor, a First-in-Class Inhibitor of Nuclear Export, in Patients With Advanced Refractory Bone or Soft Tissue Sarcoma. J Clin Oncol. 2016 Sep 10;34(26):3166-74. doi: 10.1200/JCO.2016.67.6346. Epub 2016 Jul 25. PMID 27458288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 sites in United States and Canada from 30 July 2013 to 21 October 2016.
Pre-assignment Details: A total of 54 participants were enrolled and randomized to study treatment.
Groups:
- Arm 1:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 milligrams per meter square (mg/m^2) orally twice weekly in treatment sequence ABCD (Treatment A: fasted, tablet formulation on Day 1 of Week 1; Treatment B: high-fat meal, tablet formulation on Day 1 of Week 2; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 3; Treatment D: low-fat meal, capsule formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
- Arm 2:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence BADC (Treatment B: high-fat meal, tablet formulation on Day 1 of Week 1; Treatment A: fasted, tablet formulation on Day 1 of Week 2; Treatment D: low-fat meal, capsule formulation on Day 1 of Week 3; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
- Arm 3:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 50 mg/m^2 first generation tablets twice weekly on Days 1 and 3 of each week within 30 minutes of solid food consumption.
- Arm 4:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 60 mg/m^2 orally in treatment sequence ABC (Treatment A: current [1st generation] tablets on Day 1 of Week 1; Treatment B: new [2nd generation] tablets on Day 1 of Week 2; Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
- Arm 5:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 60 mg/m^2 orally in treatment sequence CAB (Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 1; Treatment A: current [1st generation] tablets on Day 1 of Week 2; Treatment B: new [2nd generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
- Arm 6:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 60 mg/m^2 orally in treatment sequence BCA (Treatment B: new [2nd generation] tablets on Day 1 of Week 1; Treatment C: suspension dose of current [1st generation] tablets on Day 1 of Week 2; Treatment A: current [1st generation] tablets on Day 1 of Week 3 in Cycle 1 (Weeks 1 to 3). All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
Period: Overall Study
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Started | 10 | 9 | 17 | 7 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 9 | 17 | 7 | 5 | 6
Not completed — Adverse Event | 1 | 0 | 2 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 3 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1 | 0 | 0
Not completed — Disease Progression | 7 | 5 | 8 | 4 | 4 | 4
Not completed — Need of treatment not allowed per protocol | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Intercurrent illness | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least one dose of selinexor.
Groups:
- Arm 1:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence ABCD (Treatment A: fasted, tablet formulation on Day 1 of Week 1; Treatment B: high-fat meal, tablet formulation on Day 1 of Week 2; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 3; Treatment D: low-fat meal, capsule formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
- Total: Total of all reporting groups
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6: | Total
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (12.72) | 57.6 (17.18) | 59.9 (13.90) | 53.4 (8.10) | 43.6 (19.32) | 53.8 (11.62) | 55.0 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11 | 3 | 3 | 3 | 31
  Male | 6 | 2 | 6 | 4 | 2 | 3 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 7 | 16 | 7 | 4 | 6 | 49
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 1 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 2 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 0 | 3
  White | 8 | 9 | 12 | 4 | 3 | 5 | 41
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From the Time Zero to the Last Non-zero Concentration (AUC0-t) of Selinexor
Description: AUC0-t was defined as area under the concentration-time curve from time zero to the last non-zero concentration.
Time Frame: Day 1 of weeks 1-3 in Cycle 1: Pre-dose (within 10 minutes before swallowing study drug), 15, 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 10,18, 24, and 48 hours post-dose
Population: Pharmacokinetic (PK) population included all participants in Arms 1, 2 and Arms 4, 5, and 6 who received selinexor, and for whom the PK profile for all treatments could be adequately characterized. Here 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. As pre-specified in SAP and protocol Arm 3 was a non-PK group assessment, so data was not collected and analyzed for this PK outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter (ng*h/mL)
Groups:
- Arms 1 and 2: Treatment A: Fasted, Tablet Formulation: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (i.e. Treatment A: fasted, tablet formulation on Day 1 [Week 1] in Arm 1 and Day 1 [Week 2] in Arm 2).
- Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (i.e. Treatment B: high-fat meal, tablet formulation on Day 1 [Week 2] in Arm 1 and Day 1 [Week 1] in Arm 2).
- Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (i.e. Treatment C: low-fat meal, tablet formulation on Day 1 [Week 3] in Arm 1 and Day 1 [Week 4] in Arm 2).
- Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (i.e. Treatment D: low-fat meal, capsule formulation on Day 1 [Week 4] in Arm 1 and Day 1 [Week 3] in Arm 2).
- Arms 4, 5, and 6: Treatment A: First Generation Tablet: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 60 mg/m^2 orally in randomized treatment sequence (i.e. Treatment A: current [1st generation] tablets on Day 1 and 3 in Arm 4, 5 and 6 for Cycle 1 (Weeks 1 to 3).
- Arms 4, 5, and 6: Treatment B: Second Generation Tablet: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 60 mg/m^2 orally in randomized treatment sequence (i.e. Treatment B: new [2nd generation] tablets on Day 1 in Arm 4, 5 and 6 for (Weeks 1 to 3).
- Arms 4, 5, and 6: Treatment C: Oral Suspension: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 60 mg/m^2 orally in randomized treatment sequence (i.e. Treatment C: suspension dose of current [1st generation] tablets on Day 1 and 3 in Arm 4, 5 and 6 for (Weeks 1 to 3).
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Nanograms*hour per milliliter (ng*h/mL) | 2752 (37.5) | 3175 (25.3) | 3280 (19.3) | 3342 (21.4) | 4086 (22.3) | 4220 (22.0) | 3955 (21.2)

2. Primary Outcome: Area Under the Concentration Time Curve From the Time Zero to Extrapolated to Infinity (AUC0-inf) of Selinexor
Description: AUC0-inf was defined as area under the concentration-time curve from time zero to infinity (extrapolated), AUC0-inf was calculated as AUC0-t + Ct/ elimination rate constant (kel), where: Ct = the last observed non- zero concentration.
Time Frame: Day 1 of weeks 1-3 in Cycle 1: Pre-dose (within 10 minutes before swallowing study drug), 15, 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 18, 24, and 48 hours post-dose
Population: PK population included all participants in Arms 1, 2 and Arms 4, 5, and 6 who received selinexor, and for whom the PK profile for all treatments could be adequately characterized. Here 'overall number of participants analyzed' signifies participants who are evaluable for this outcome measure. As pre-specified in SAP and protocol Arm 3 was a non-PK group assessment, so data was not collected and analyzed for this PK outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
ng*h/mL | 2969 (34.1) | 3412 (23.8) | 3483 (18.1) | 3561 (20.6) | 4117 (22.4) | 4250 (21.8) | 4002 (21.1)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Selinexor
Description: Cmax was defined as maximum observed concentration, taken directly from the plasma concentration data.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Nanogram per milliliter (ng/mL) | 355 (52.6) | 404 (39.1) | 436 (21.9) | 429 (29.1) | 519 (34.4) | 527 (30.7) | 450 (52.8)

4. Primary Outcome: Time of First Maximum Observed Concentration (Tmax) of Selinexor
Description: Tmax was defined as time of first observation of Cmax, taken directly from the plasma concentration data.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Groups:
- Arms 1 and 2: Treatment A: Fasted, Tablet Formulation: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received Selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (i.e. (i.e. Treatment A: fasted, tablet formulation on Day 1 [Week 1] in Arm 1 and Day 1 [Week 2] in Arm 2).
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Hour | 1.5 [1.0 to 6.1] | 3.4 [1.5 to 8.0] | 3.4 [1.4 to 6.1] | 3.8 [1.5 to 5.0] | 2.1 [0.6 to 5.1] | 3.0 [1.0 to 4.2] | 1.6 [1.0 to 9.7]

5. Primary Outcome: Terminal Phase Half-Life (t1/2) of Selinexor
Description: t1/2 was the terminal phase half-life, it was calculated as ln(2)/kel.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Groups:
- Arms 4, 5, and 6: Treatment A: First Generation Tablet: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 60 mg/m^2 orally in randomized treatment sequence (i.e. Treatment A: current [1st generation] tablets on Day 1 and 3 [Week 1 and 3] in Arm 4 and 6 and Day 1 [Week 2] in Arm 2 for one cycle (Weeks 1 to 3).
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Hour | 6.2 (1.71) | 5.9 (1.36) | 5.6 (1.00) | 5.7 (1.06) | 6.7 (1.34) | 6.6 (1.14) | 6.5 (1.51)

6. Primary Outcome: Apparent Total Body Clearance (CL/F) of Selinexor
Description: Apparent total body clearance was calculated as Dose/AUC0-inf, uncorrected for fraction absorbed; reported normalized by participant body weight (kilogram [kg]).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour per kilogram (L/h/kg)
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Liter per hour per kilogram (L/h/kg) | 0.3 (32.1) | 0.22 (21.3) | 0.22 (16.3) | 0.21 (18.7) | 0.21 (20.6) | 0.20 (16.6) | 0.21 (14.2)

7. Primary Outcome: Apparent Volume of Distribution (Vd/F) of Selinexor
Description: Vd/F was calculated as Dose/ (kel *AUC0-inf), uncorrected for fraction absorbed; reported normalized by participant body weight (kg).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per kilogram (L/kg)
Arm/Group | Arms 1 and 2: Treatment A: Fasted, Tablet Formulation | Arms 1 and 2: Treatment B: High-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment C: Low-Fat Meal, Tablet Formulation | Arms 1 and 2: Treatment D: Low-Fat Meal, Capsule Formulation | Arms 4, 5, and 6: Treatment A: First Generation Tablet | Arms 4, 5, and 6: Treatment B: Second Generation Tablet | Arms 4, 5, and 6: Treatment C: Oral Suspension
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 13 | 13
Liter per kilogram (L/kg) | 2.2 (49.5) | 1.8 (32.3) | 1.7 (26.1) | 1.7 (26.6) | 2.0 (16.9) | 1.9 (18.3) | 1.9 (18.2)

8. Secondary Outcome: Percentage of Participants With Best Overall Response According to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 Criteria
Description: Best overall response rate was defined as the percentage of participants who achieved complete response (CR), and partial response (PR), as assessed by the RECIST v1.1 criteria. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non target) must have reduction in the short axis to less than (<) 10 millimeter (mm). PR was defined as At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameter (LD).
Time Frame: From the date of first documented response until the date of documented progression or last disease assessment (up to 39 months)
Population: Safety population consisted of all participants who received at least one dose of selinexor. Data for this outcome measure analysis was planned to be analyzed as per disease specific sarcoma.
Measure: Number; unit: Percentage of participants
Groups:
- Liposarcoma: Participants with liposarcoma received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (A, B, C, D) in Arm 1 and 2 for one cycle (Weeks 1 to 4); 50 mg/m^2 first generation tablets twice weekly on Days 1 and 3 in Arm 3; 60 mg/m^2 orally in randomized treatment sequence (A, B, C) on Day 1 and 3 for 1st generation tablets and Day 1 for 2nd generation tablets for one cycle (Weeks 1 to 3).
- Leiomyosarcoma: Participants with leiomyosarcoma received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (A, B, C, D) in Arm 1 and 2 for one cycle (Weeks 1 to 4); 50 mg/m^2 first generation tablets twice weekly on Days 1 and 3 in Arm 3; 60 mg/m^2 orally in randomized treatment sequence (A, B, C) on Day 1 and 3 for 1st generation tablets and Day 1 for 2nd generation tablets for one cycle (Weeks 1 to 3).
- Other Sarcoma: Participants with Other sarcoma received selinexor 30 mg/m^2 orally twice weekly in randomized treatment sequence (A, B, C, D) in Arm 1 and 2 for one cycle (Weeks 1 to 4); 50 mg/m^2 first generation tablets twice weekly on Days 1 and 3 in Arm 3; 60 mg/m^2 orally in randomized treatment sequence (A, B, C) on Day 1 and 3 for 1st generation tablets and Day 1 for 2nd generation tablets for one cycle (Weeks 1 to 3).
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 19 | 12 | 23
Percentage of participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0

9. Secondary Outcome: Duration of Stable Disease as Per RECIST v1.1 Criteria
Description: Duration of at least stable disease was defined as the time from the date of first dose of study treatment to first documented radiologic evidence of disease recurrence or progression as per RECIST v1.1 Criteria. Participants without evidence of progression were censored at time of last disease assessment. Progressive Disease (PD) was defined as at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded since the treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions also constituted progressive disease.
Time Frame: From the date of first dose of study treatment to first documented radiologic evidence of disease recurrence or progression, censored date (up to 39 months)
Population: Safety population consisted of all participants who received at least one dose of selinexor. Data for this outcome measure was planned to be analyzed as per disease specific sarcoma.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 19 | 12 | 23
Months | 7.49 [3.55 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 3.94 [1.64 to 5.55] | 8.34 [3.09 to NA] — Data could not be estimated due to higher number (>50%) of censored participants.

10. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST v1.1 Criteria
Description: PFS was defined as the time from the date of randomization until the first date of Independent Review Committee (IRC)-confirmed PD per RECIST v1.1, or death due to any cause. PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest sum of the longest diameter (SLD) recorded from baseline or the appearance of 1 or more new lesions. Participants who were last known to be alive and without evidence of progression were censored at time of last disease assessment. If date of progression or death occurred after more than 1 missed disease assessment interval, or 30 days after end of treatment, participants were censored at the time of last evaluable disease assessment prior to the missed assessment.
Time Frame: From first dose of study treatment to time of disease progression or death, censored date (up to 39 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 19 | 12 | 23
Months | 4.44 [2.07 to 7.49] | 3.52 [1.48 to 5.55] | 1.84 [1.02 to 3.58]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date first dose of study treatment to the date of death. Participants who were still alive prior to the data cutoff for final efficacy analysis, or who dropped out prior to study end, were censored at the day they were last known to be alive.
Time Frame: From first dose of study treatment to death, censored date (up to 39 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 19 | 12 | 23
Months | 9.00 [4.76 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 7.03 [5.75 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | NA [3.38 to NA] — Data could not be estimated due to higher number (>50%) of censored participants.

12. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from date of first dose of study treatment to first documented evidence of disease recurrence or progression, or death due to disease progression, whichever occurred first. Participants without evidence of progression were censored at time of last evaluable disease assessment.
Time Frame: From first dose of study treatment to first documented evidence of disease recurrence or progression, or death, censored date (up to 39 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 19 | 12 | 23
Months | 4.44 [2.07 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 3.52 [1.48 to 5.55] | 1.74 [1.02 to 5.55]

13. Secondary Outcome: Number of Participants With Growth Modulation Index (GMI) Less Than or Equal to (<=) 1.33 and Greater Than (>) 1.33
Description: GMI was defined as the ratio between the TTP with selinexor and the TTP with the most recent prior treatment. GMI was calculated, using a previously described threshold of 1.3 or greater as a sign of potential drug activity and improved overall survival.
Time Frame: Up to 39 months
Population: Safety population consisted of all participants who received at least one dose of selinexor. Data for this outcome measure was planned to be analyzed as per disease specific sarcoma. Here 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposarcoma | Leiomyosarcoma | Other Sarcoma
Number analyzed (Participants) | 18 | 12 | 20
Participants
  GMI <= 1.33 | 11 | 8 | 17
  GMI > 1.33 | 7 | 4 | 3

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a study and which does not necessarily have to have a causal relationship with this treatment. SAE defined as any AE, occurring at any dose (including after the informed consent form was signed and prior to dosing) that and regardless of causality that: results in death, is life-threatening (participant was at immediate risk of death from event as it occurred), requires in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect. TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study treatment through 30 days following last dose or any event considered drug-related by the investigator through the end of the study.
Time Frame: From screening up to 30 days post last study drug dose (up to 39 months)
Population: Safety population consisted of all participants who received at least one dose of selinexor. As pre-specified in SAP, safety data was collected and analyzed as per the individual arms with specified treatment sequences only.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence BADC (Treatment B: high-fat meal, tablet formulation on Day 1 of Week 1; Treatment A: fasted, tablet formulation on Day 1 of Week 2; Treatment D: lowfat meal, capsule formulation on Day 1 of Week 3; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6
Participants
  Participants with TEAEs | 10 | 9 | 17 | 7 | 5 | 6
  Participants with Serious TEAEs | 4 | 5 | 5 | 2 | 2 | 4

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: AE was defined as the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition that occur after participant's signed informed consent obtained. TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study treatment through 28 days following last dose or any event considered drug-related by the investigator through the end of the study. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death.
Time Frame: From screening up to 30 days post last study drug dose (up to 39 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence BADC (Treatment B: high-fat meal, tablet formulation on Day 1 of Week 1; Treatment A: fasted, tablet formulation on Day 1 of Week 2; Treatment D: low fat meal, capsule formulation on Day 1 of Week 3; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6
Participants
  Grade 1: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2: Moderate | 3 | 2 | 2 | 1 | 1 | 1
  Grade 3: Severe | 5 | 5 | 14 | 3 | 2 | 4
  Grade 4: Life Threatening | 2 | 1 | 0 | 3 | 1 | 1
  Grade 5: Fatal | 0 | 1 | 1 | 0 | 1 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Number of participants with clinically significant laboratory abnormalities including clinical chemistry, hematology, coagulation and urinalysis. Number of participants with clinically significant laboratory abnormalities which were deemed clinically significant by the investigator were reported.
Time Frame: From screening up to 30 days post last study drug dose (up to 39 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6
Participants
  Hematology | 1 | 2 | 7 | 1 | 2 | 1
  Clinical Chemistry | 4 | 1 | 7 | 1 | 1 | 1
  Coagulation: Prothrombin intl. normalized ratio | 0 | 0 | 1 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included blood pressure (systolic blood pressure and diastolic blood pressure). Measurements were made after the participant had been resting supine for a minimum of 5 minutes. Clinically significant findings were defined as such in the opinion of the investigator occurring at any time on treatment from normal pre-dose based on the condition met (Yes/No). Number of participants with clinically significant changes in vital signs with condition (Yes) were only reported.
Time Frame: From screening up to 30 days post last study drug dose (up to 39 months)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6
Participants
  Systolic Blood Pressure: < 100 mmHg (Yes) | 2 | 5 | 8 | 4 | 3 | 3
  Systolic Blood Pressure: > 10 mmHg decrease from baseline (Yes) | 3 | 7 | 14 | 6 | 5 | 5
  Systolic Blood Pressure: > 20 mmHg decrease from baseline (Yes) | 2 | 4 | 10 | 4 | 1 | 3
  Systolic Blood Pressure: < 100 mmHg and > 10 mmHg decrease from baseline (Yes) | 1 | 4 | 7 | 3 | 3 | 2
  Systolic Blood Pressure: < 100 mmHg and > 20 mmHg decrease from baseline (Yes) | 1 | 1 | 4 | 2 | 1 | 2
  Diastolic Blood Pressure: < 60 mmHg (Yes) | 2 | 3 | 10 | 2 | 2 | 2
  Diastolic Blood Pressure: > 5 mmHg decrease from baseline (Yes) | 8 | 7 | 15 | 6 | 4 | 5
  Diastolic Blood Pressure: > 10 mmHg decrease from baseline (Yes) | 5 | 5 | 12 | 5 | 3 | 4
  Diastolic Blood Pressure: < 60 mmHg and > 5 mmHg decrease from baseline (Yes) | 2 | 2 | 9 | 2 | 1 | 2
  Diastolic Blood Pressure: < 60 mmHg and > 10 mmHg decrease from baseline (Yes) | 2 | 2 | 9 | 2 | 0 | 2
  Systolic Blood Pressure : > 140 mmHg (Yes) | 2 | 3 | 6 | 2 | 3 | 3
  Systolic Blood Pressure: > 160 mmHg (Yes) | 0 | 0 | 1 | 1 | 0 | 0
  Systolic Blood Pressure: > 10 mmHg increase from baseline (Yes) | 2 | 6 | 11 | 3 | 4 | 5
  Systolic Blood Pressure: > 20 mmHg increase from baseline (Yes) | 1 | 5 | 3 | 1 | 1 | 4
  Systolic Blood Pressure: > 160 mmHg and > 10 mmHg increase from baseline (Yes) | 0 | 0 | 1 | 1 | 0 | 0
  Systolic Blood Pressure: > 160 mmHg and > 20 mmHg increase from baseline (Yes) | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure: > 90 mmHg (Yes) | 4 | 3 | 6 | 2 | 3 | 3
  Diastolic Blood Pressure: > 100 mmHg (Yes) | 0 | 0 | 1 | 1 | 0 | 0
  Diastolic Blood Pressure: > 5 mmHg increase from baseline (Yes) | 6 | 5 | 13 | 4 | 4 | 6
  Diastolic Blood Pressure: > 10 mmHg increase from baseline (Yes) | 2 | 4 | 8 | 2 | 3 | 4
  Diastolic Blood Pressure: > 100 mmHg and > 5 mmHg increase from baseline (Yes) | 0 | 0 | 1 | 1 | 0 | 0
  Diastolic Blood Pressure: > 100 mmHg and > 10 mmHg increase from baseline (Yes) | 0 | 0 | 0 | 1 | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECGs)
Description: Twelve lead ECGs were obtained after the participant has rested in a supine position for at least 5 minutes. Clinically significant findings were defined as such in the opinion of the investigator or designated physician occurring at any time on treatment from normal pre-dose.
Time Frame: From screening up to 30 days post last study drug dose
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
Number analyzed (Participants) | 10 | 9 | 17 | 7 | 5 | 6
Participants | 2 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to 30 days post last study drug dose (up to 39 months)
Description: Safety population consisted of all participants who received at least one dose of selinexor. As pre-specified in SAP, safety data was collected and analyzed as per the individual arms with specified treatment sequences only.
Groups:
- Arm 2:: Participants with advanced sarcomas (Liposarcoma, Leiomyosarcoma, and Other sarcoma) received selinexor 30 mg/m^2 orally twice weekly in treatment sequence BADC (Treatment B: high-fat meal, tablet formulation on Day 1 of Week 1; Treatment A: fasted, tablet formulation on Day 1 of Week 2; Treatment D: low fat meal, capsule formulation on Day 1 of Week 3; Treatment C: low-fat meal, tablet formulation on Day 1 of Week 4 in Cycle 1 (Weeks 1 to 4).All participants received the current (1st generation) tablet formula at a dose of 60 mg on Day 3 of Weeks 1-3 of Cycle 1.
Arm/Group | Arm 1: | Arm 2: | Arm 3: | Arm 4: | Arm 5: | Arm 6:
All-Cause Mortality (participants affected / at risk) | 2/10 | 2/9 | 1/17 | 3/7 | 3/5 | 2/6
Serious Adverse Events (participants affected / at risk) | 4/10 | 5/9 | 5/17 | 2/7 | 2/5 | 4/6
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 17/17 | 7/7 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: (N=10) | Arm 2: (N=9) | Arm 3: (N=17) | Arm 4: (N=7) | Arm 5: (N=5) | Arm 6: (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: (N=10) | Arm 2: (N=9) | Arm 3: (N=17) | Arm 4: (N=7) | Arm 5: (N=5) | Arm 6: (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 12 | 1 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 8 | 9 | 1 | 5 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 7 | 6 | 0 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 5 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Left atrial enlargement (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 8 | 1 | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 2 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 17 | 6 | 4 | 5
Constipation (Gastrointestinal disorders) | 5 | 5 | 12 | 3 | 2 | 5
Vomiting (Gastrointestinal disorders) | 5 | 5 | 12 | 4 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 5 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 8 | 9 | 16 | 4 | 5 | 6
Oedema peripheral (General disorders) | 3 | 2 | 4 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 4 | 0 | 2 | 0
Chills (General disorders) | 2 | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Face oedema (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Cement embolism (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 3 | 8 | 2 | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 1 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 2 | 1 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 2 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 10 | 4 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5 | 6 | 3 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 5 | 0 | 2 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 1 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 2 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 5 | 8 | 0 | 1 | 4
Dizziness (Nervous system disorders) | 2 | 3 | 11 | 1 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 4 | 2 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 3 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 2 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 7 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 8 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nail cuticle fissure (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 3 | 1 | 3 | 1
Hypertension (Vascular disorders) | 1 | 1 | 4 | 2 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other